CLINICAL TRIAL: NCT04690322
Title: POCUS: Hemostatic Potential and Joint Health in Patients With Severe Hemophilia A on Novel Replacement Therapies
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Garcia, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-1378
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia A; Factor VIII
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein; BAX 855; emicizumab; Solutions

STUDY DESIGN:
Intervention Model Description: Each patient will be randomly assigned to receive either extended half-life factor VIII based replacement therapy or non-FVIII based replacement therapy
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Extended half-life factor VIII-based replacement therapy (Active Comparator): Subjects who are either already on prophylactic standard half-life FVIII products or have not started prophylactic treatment will be randomized to start prophylactic extended half-life FVIII products or non-factor product (emicizumab). Both therapies are considered the current standard of care.
  The study has 4 planned visits at baseline, 1 month, 6 months, and 12 months. They will coincide with the standard of care visits.
  Interventions: Drug: Eloctate; Drug: Adynovate
- Non-Factor VIII-based replacement therapy (Active Comparator): Subjects who are either already on prophylactic standard half-life FVIII products or have not started prophylactic treatment will be randomized to start prophylactic extended half-life FVIII products or non-factor product (emicizumab). Both therapies are considered the current standard of care.
  The study has 4 planned visits at baseline, 1 month, 6 months, and 12 months. They will coincide with the standard of care visits.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Eloctate — Eloctate is FDA-approved to treat patients with Hemophilia A. This drug will be used for extended half-life factor VIII-based replacement therapy.
  Other Names: ELOCTATE- antihemophilic factor (recombinant), fc fusion protein
  Arms: Extended half-life factor VIII-based replacement therapy
Drug: Adynovate — Adynovate is FDA-approved to treat patients with Hemophilia A. This drug will be used for extended half-life factor VIII-based replacement therapy.
  Other Names: ADYNOVATE- antihemophilic factor (recombinant) pegylated
  Arms: Extended half-life factor VIII-based replacement therapy
Drug: Emicizumab — Emicizumab is FDA-approved to treat patients with Hemophilia A. This drug will be used for non-factor VIII-based replacement therapy.
  Other Names: HEMLIBRA- emicizumab injection, solution
  Arms: Non-Factor VIII-based replacement therapy

SUMMARY:
This is a prospective, randomized control trial in which each patient will be randomly assigned to receive either extended half-life factor VIII based replacement therapy or non-FVIII based replacement therapy, which are both standard of care treatment for persons with Hemophilia A.

DETAILED DESCRIPTION:
This is a research study to find out if there is a difference in the way children with hemophilia A form a clot and also evaluate if they develop tiny bleeds within the joint and subsequently early joint changes when receiving extended half-life factor VIII based replacement therapy vs non-FVIII based replacement as part of their hemophilia treatment to prevent spontaneous joint bleeds.

Both therapies are standard of care therapies for patients with hemophilia A. The only experimental/research procedures as part of this study include the thrombin generation assay and ultrasound. All other procedures are standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate hemophilia A (baseline factor VIII activity 1-5%) or severe hemophilia A (baseline factor VIII activity <1%) on prophylactic standard half-life FVIII infusions OR subjects with moderate or severe hemophilia A who have not started prophylactic treatment
* Less than 18 years of age

Exclusion Criteria:

* Subjects with documented FVIII inhibitor
* Subjects with a history of ≥ 2 target joints
* Subjects with a history of synovectomy
* Currently using medications known to impact bone and mineral metabolism (e.g., bisphosphonates, corticosteroids, estrogen, testosterone, calcitonin, thyroid hormone therapy);
* Disease states known to affect bone integrity (e.g., primary hyperparathyroidism, Paget's disease, clinically significant liver disease)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Changes in hemostatic potential | Baseline, 1 month, 6 months, and 12 months from start of study
  Evaluate differences in hemostatic potential in persons with hemophilia A without evidence of hemophilic target joints who are receiving prophylactic FVIII-based replacement therapy versus non-FVIII replacement therapy by measuring thrombin generation potential via a plasma-based assay
Changes in early joint-health markers | Baseline, 1 month, 6 months, and 12 months from the start of study
  Identify early joint-health markers associated with bleeding in persons with hemophilia A without evidence of hemophilic target joints who are receiving prophylactic FVIII-based replacement therapy versus non-FVIII replacement by measuring soft tissue and osteochondral changes among 6 joints (bilateral elbows, knees, and ankles) using point of care ultrasound between both treatment groups

SECONDARY OUTCOMES:
Changes in bleeding rates | Baseline and 12 months after start of study
  Measure bleeding rates in persons with hemophilia A without evidence of hemophilic target joints on prophylactic FVIII-based replacement therapy versus non-FVIII replacement therapy by measuring the difference in annualized bleeding rates between the two treatment groups, as well as other surrogate markers of bleeding, or indirect causes of bleeding, which include FVIII inhibitor level, hemoglobin, and serum ferritin
Changes in health-related quality of life and physical activity | Baseline, 1 month, 6 months, and 12 months from the start of study
  Evaluate health-related quality of life and physical activity in persons with hemophilia A without evidence of hemophilic target joints on prophylactic FVIII-based replacement therapy versus non-FVIII replacement therapy using validated questionnaires
Changes in joint health | Baseline, 1 month, 6 months, and 12 months from the start of study
  Assess joint health in persons with hemophilia A without evidence of hemophilic target joints on prophylactic FVIII-based replacement therapy versus non-FVIII replacement therapy using validated outcome tool (Hemophilia Joint Health Score)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Garcia, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States